CLINICAL TRIAL: NCT05965492
Title: Optimal Multimodal Pain Management Package Versus Regular Bottled Pain Formulation for Outpatient Use Following Microdiscectomies , Foraminotomies, and Spinal Decompressions: A Randomized Control Trial Comparing Two Strategies
Brief Title: Multimodal Pain Package vs. Regular Formulation for Pain Management in Ambulatory Spinal Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study drug was not compliant with research pharmacy
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Yiliam Rodriguez, Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230423
Record Dates: First submitted 2023-07-12; First posted 2023-07-28 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Spinal Disorder
MeSH Terms: conditions — Spinal Diseases | interventions — Acetaminophen; Celecoxib; Gabapentin; Famotidine; Calcium Dobesilate; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bottled pain formulations Group (Active Comparator): Participants in this group will use the standard-of-care medication treatment for ambulatory spinal surgery prescribed to them in different bottles for 7 days.
  Interventions: Drug: Acetaminophen; Drug: Celebrex; Drug: Gabapentin; Drug: Famotidine; Drug: Decadron; Drug: Oxycodone
- Multi-Modal regimen Group (Experimental): Participants in this group will receive the same drugs used during the standard-of-care treatment for ambulatory spinal surgery. However, the drugs will be prescribed using a simple multimodal medication pre-formulated package for 7 days.
  Interventions: Drug: Acetaminophen; Drug: Celebrex; Drug: Gabapentin; Drug: Famotidine; Drug: Decadron; Drug: Oxycodone

INTERVENTIONS:
Drug: Acetaminophen — Day 1 and Day 2: 1000 mg three times a day administered via tablet by mouth for a total cumulative daily dose of 3000 mg.
  Day 3 and Day 4: 825 mg three times a day administered via tablet by mouth for a total cumulative daily dose of 2475 mg.
  Day 5: 500 mg two times a day and 325 mg once a day administered via tablet by mouth for a total cumulative daily dose of 1325 mg.
  Day 6: 500 mg once a day and 325mg twice a day administered via tablet by mouth for a total cumulative daily dose of 1150 mg.
  Day 7: 500 mg twice a day administered via tablet by mouth for a total cumulative daily dose of 1000 mg.
Drug: Celebrex — Day 1: 200 mg twice a day administered via tablet by mouth for a total cumulative daily dose of 400 mg.
  Day 2 and Day 3: 100 mg three times a day administered via tablet by mouth for a total cumulative daily dose of 300 mg.
  Day 4: 100 mg twice a day administered via tablet by mouth for a total cumulative daily dose of 200 mg.
  Day 5: 50 mg twice a day administered via tablet by mouth for a total cumulative daily dose of 100 mg.
  Not prescribed on Days 6 and 7.
Drug: Gabapentin — Day 1 and Day 2: 300 mg three times a day administered via tablet by mouth for a total cumulative daily dose of 900 mg.
  Day 3: 200 mg three times a day administered via tablet by mouth for a total cumulative daily dose of 600 mg.
  Day 4: 200 mg two times a day and 100mg once a day administered via tablet by mouth for a total cumulative daily dose of 500 mg.
  Day 5: 100 mg three times a day administered via tablet by mouth for a total cumulative daily dose of 300 mg.
  Day 6: 100 mg two times a day administered via tablet by mouth for a total cumulative daily dose of 200 mg.
  Day 7: 100 mg once a day administered via tablet by mouth for a total cumulative daily dose of 100 mg.
Drug: Famotidine — Day 1- Day 7: 20 mg once a day administered via tablet by mouth for a total cumulative daily dose of 20 mg.
Drug: Decadron — Day 1: 4 mg three times a day administered via tablet by mouth for a total cumulative daily dose of 12 mg.
  Day 2: 4 mg two times a day administered via tablet by mouth for a total cumulative daily dose of 8 mg.
  Day 3: 2 mg two times a day administered via tablet by mouth for a total cumulative daily dose of 4 mg.
  Not prescribed on Days 4 through 7.
Drug: Oxycodone — A prescription of oxycodone as per standard of care will be provided to participants in case of breakthrough pain.

SUMMARY:
The purpose of this research is to compare two outpatient pain management strategies in patients undergoing spinal surgeries such as microdiscectomies, foraminotomies, and spinal decompressions.

ELIGIBILITY:
Inclusion Criteria:

* Adults: males or non-pregnant females.
* Patients undergoing ambulatory microdiscectomies, foraminotomies, and spinal cord decompressions requiring pain control analgesics.

Exclusion Criteria:

* Pregnancy
* Active severe liver disease
* Chronic kidney disease 3a-5 (moderate to severe)
* Chronic obstructive pulmonary disease with impaired pulmonary function
* Chronic steroid use
* Chronic opioid use
* Current use of narcotics
* Allergy to sulfonamides
* Allergy to NSAIDs
* Allergy to Aspirin
* Allergy to Tylenol
* Allergy to Gabapentins
* Allergy to H2 blockers (cimetidine, famotidine)
* Allergy to steroid
* Current use of gabapentins for any medical condition
* Inability to be discharged home on the day of surgery
* Inability to swallow pills
* Myasthenia gravis
* History of gastrointestinal ulcers or stomach bleeding
* Have any condition that, in the investigator's opinion, will compromise the well-being of the patient or the study, or prevent the patient from meeting or performing study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Adherence measured by the self-report medication nonadherence scale | up to 7 days
  Adherence will be measured using a Likert scale ranging from "never" indicating that the participant followed all instructions and adhered to the medication to "all the time. "indicating that the participant never followed instructions and did not take the medication.
Satisfaction measured by Satisfaction Likert Scale | up to 7 days
  Scores range from "0" not satisfied to "10" very satisfied
Ease of use as measured by Likert Scale | up to 7 days
  Scores ranges from "strongly disagree to Strongly agree" regarding the ease of use of the medication package.

SECONDARY OUTCOMES:
Number of pain pills | up to 7 days
  Count of pills taken by participants

CONTACTS AND LOCATIONS:
Overall Officials: Yiliam Yiliam, MD, Principal Investigator — Professor of Clinical

IPD SHARING:
Plan to Share IPD: No